CLINICAL TRIAL: NCT07142733
Title: Inducing and Relieving Factors of Chest Tightness (Pain) in Patients With Acute Coronary Syndrome
Acronym: ACS
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202402091RIND
Record Dates: First submitted 2025-07-16; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2024-03

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The research aims to investigate various aspects related to chest discomfort (pain) in patients diagnosed with Acute Coronary Syndrome (ACS). Firstly, it seeks to identify the factors that trigger such discomfort in ACS patients. Additionally, the study aims to explore different methods utilized to alleviate chest pain in these individuals and assess their effectiveness. Furthermore, it aims to analyze how basic attributes of patients may influence both the precipitating factors and the effectiveness of relief methods for chest discomfort. Finally, the research aims to understand how factors related to other diseases may impact chest discomfort and its alleviation methods in ACS patients.

DETAILED DESCRIPTION:
The inclusion criteria for this study comprise patients aged 18 years or older who are proficient in communicating with the researcher in Mandarin or Taiwanese Hokkien. Exclusion criteria include individuals currently diagnosed with a mental illness, those with substance abuse or alcohol addiction, and those experiencing acute onset symptoms without a prior history of chest discomfort or pain related to heart issues.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for this study comprise patients aged 18 years or older who are proficient in communicating with the researcher in Mandarin or Taiwanese Hokkien.

Exclusion Criteria:

* Exclusion criteria include individuals currently diagnosed with a mental illness, those with substance abuse or alcohol addiction, and those experiencing acute onset symptoms without a prior history of chest discomfort or pain related to heart issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome presenting with chief complaints of chest tightness or pain.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Inducing and Relieving Factors of Chest Tightness (Pain) in Patients with Acute Coronary Syndrome | after 142 case
  The finding of this study can be used as a reference for inducing factors and relieving factors in patient with ACS.

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Li Kao, Study Chair — manager and staff
Locations (1):
- Republic of China, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided